CLINICAL TRIAL: NCT06155760
Title: Role of Extended Low Dose Prednisolone in Achieving Clinical and Biochemical Remission in Steroid Responsive Severe Alcoholic Hepatitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALD-03
Record Dates: First submitted 2023-11-16; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-10

CONDITIONS: Severe Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Steroid Therapy (Experimental): 10mg of prednisolone plus standard medical therapy for 60 days. SMT- IV Albumin, Diuretics, Multi vitamins as per clinicians decision
  Interventions: Drug: Prednisolone; Other: Standard Medical therapy
- Placebo group (Active Comparator): Standard treatment plus placebo that the patient would receive included in the trial.
  SMT- IV Albumin, Diuretics, Multi vitamins as per clinicians decision
  Interventions: Other: Standard Medical therapy; Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — 10mg of prednisolone plus standard medical therapy for 60 days
  Arms: Extended Steroid Therapy
Other: Standard Medical therapy — IV Albumin, Diuretics, Multi vitamins as per clinicians decision
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
Severity of alcoholic hepatitis is defined by Maddrey's discriminant function, value of 32 or higher indicates severe alcoholic hepatitis that carries an adverse prognosis with one month mortality of 30%-50%. Prednisolone (40 mg/day) given orally should be considered to improve 28-day mortality in patients with severe AH. Abstinence is key to long-term survival.

According to current protocol, we discontinue the treatment after 28 days but only 15 % patient is achieving the DF < 32 after 28 days of treatment.

The aim of this study is to evaluate the role of extended low dose prednisolone (10mg) in achieving remission by day-90 in steroid responsive severe alcoholic hepatitis.

DETAILED DESCRIPTION:
Study Design- Single center, Open label, Randomized controlled trial

* According to current protocol, we discontinue the treatment after 28 days, it improve the mortality rate in severe alcoholic patient with mDF score of more than 32 but only 15% patient is achieving the mDF < 32 after 28 days of treatment.
* Abstinence is key to long-term survival. No data is available in giving steroids for more than 28days going to improve clinical or biochemical parameter of the patient.

Methodology:

* Study population: All patients aged ≥ 18 years and ≤ 60 years admitted in Institute of Liver and Biliary Sciences, New Delhi with Severe Alcoholic hepatitis mDF of more than 32 days after 28days of steroid therapy and are giving written consent for participation in the study. Option of LDLT, Plasma exchange, FMT, GM- CSF given to patient with DF more than 32 after 28 days of steroid therapy and these patients are excluded from the study.
* Study period - 1.5 years after IEC approval
* Sample size - We are enrolling 150 patients.- Assuming that the response rate is 50% in prednisolone + SMT group and 20% in only SMT group. With alpha- 5% and power of 80, we need to enroll - 90 cases i.e, 45 in each group. Further adding 10% drop out cases, it was decided to enroll 100 patients i.e, 50 in each group. Allocation will be done randomly by block randomization panel by block size of 10. Further assuming that DF > 32 will be in 80% cases we need to enroll 125 cases. Further 80% will have lille score < 0.45, so it is to decide to enroll 150 cases.
* Intervention - Extended steroid group: 10mg of prednisolone plus standard medical therapy for 60 days.
* Placebo group: Standard treatment plus placebo that the patient would receive included in the trial.
* SMT- IV Albumin, Diuretics, Multi vitamins as per clinicians decision
* Monitoring and assessment:
* Investigations - Tests performed on Day 0, 4, 7, 28, 60 and 90.

  * Routine: CBC, RFT, LFT, PT/INR, CXR, PCT, Urine R/M & C/S, Blood C/S,
  * Blood sugar- fasting & PP.
* Statistical Analysis: The data will be represented as mean ± SD. The categorical data will be analysed using Chi-square test. The continuous data will be analysed by student T test, or Mann-Whitney test, whichever is applicable. Besides this, Cox regression will be applied to analyse the variables. For all tests, p≤ 0.05 will be considered statistically significant
* Adverse effects
* New onset Diabetes, risk of infection
* Stopping rule
* Discontinuation of steroids (variceal bleed, infections, uncontrolled sugars, new onset AKI)
* Death
* Liver transplantation
* Lapse or relapse of alcohol consumption

Expected outcome of the project:

- Improvement in the mDF score (<32) i.e. Remission in severe alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Persistence of mDF > 32 at day 28 of steroids.

Exclusion Criteria:

1. Active infection
2. Uncontrolled sugars
3. No consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
To assess the proportion of steroid responsive SAH patients achieving remission by extended low dose Prednisolone (10mg/day) till day 90 in comparison to SMT | 90 days

SECONDARY OUTCOMES:
Changes in the liver disease severity parameters like CTP, MELD-Na, DF, by extending the low dose steroids by 2 months in the study group compared with the control group. | 90 days
Number of patients with SAH achieving 90 day transplant-free survival between the two groups. | 90 day, 180 day
New onset infections, diabetes | 90 days
  To check new onset of infection as suspected by clinical presentation and by laboratory tests such as procalcitonin, Urine Culture, Blood Culture, chest X- Ray and Ascitic fluid analysis. And for measuring diabetes onset regular fasting and post prandial sugar charting on weekly basis throughout the study period.
90 day readmission rates | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided